CLINICAL TRIAL: NCT07078500
Title: A Prospective, Single-Arm, Multicenter Clinical Study of Orelabrutinib Combined With Pola-R-CHP Regimen for the Treatment of Untreated Non-GCB Diffuse Large B-Cell Lymphoma
Brief Title: Orelabrutinib Combined With Pola-R-CHP Regimen for the Treatment of Untreated Non-GCB Diffuse Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Second Affiliated Hospital of Jiaxing University (Other); Taizhou First People's Hospital (Other); Huzhou Central Hospital (Other); Zhejiang Cancer Hospital (Other); Dongyang People's Hospital (Other); Yuyao People's Hospital (Other); Taizhou Hospital (Other); Shaoxing Central Hospital (Other); Affiliated Hospital of Jiaxing University (Other); Shaoxing People's Hospital (Other); The Central Hospital of Lishui City (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Ningbo People's Hospital (Unknown); The People's Hospital of Quzhou (Other); Zhuji People's hospital (Unknown); Affiliated Hangzhou First People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0086
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-02

CONDITIONS: Diffuse Large B-Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- orelabrutinib combined with the Pola-R-CHP regimen (Experimental): Enrolled patients will receive six cycles of orelabrutinib in combination with the Pola-R-CHP regimen, with each 21-day period being one cycle. At the end of the six cycles, an interim efficacy evaluation will be conducted. Patients with a response of CR or PR will receive an additional two cycles of orelabrutinib in combination with rituximab and undergo a final efficacy evaluation. Patients with a response of CR/PR after eight cycles of induction therapy will receive maintenance treatment with orelabrutinib for up to two years.
  Interventions: Drug: orelabrutinib combined with the Pola-R-CHP regimen

INTERVENTIONS:
Drug: orelabrutinib combined with the Pola-R-CHP regimen — Enrolled patients will receive six cycles of orelabrutinib in combination with the Pola-R-CHP regimen, with each 21-day period being one cycle. At the end of the six cycles, an interim efficacy evaluation will be conducted. Patients with a response of CR or PR will receive an additional two cycles of orelabrutinib in combination with rituximab and undergo a final efficacy evaluation. Patients with a response of CR/PR after eight cycles of induction therapy will receive maintenance treatment with orelabrutinib for up to two years.

SUMMARY:
Assess the preliminary efficacy and safety of orelabrutinib in combination with the Pola-R-CHP regimen for the treatment of treatment-naive Non-GCB diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Currently, the R-CHOP regimen can cure approximately 60% of DLBCL patients. The Pola-R-CHP regimen has shown further improvement on this basis. However, from the POLARIX study, it was observed that patients under 60 years old, with an IPI score of 2, and those with large masses did not show further benefits from the Pola regimen. Meanwhile, for patients with poor prognosis such as non-GCB, there is still room for further improvement with the Pola-R-CHP regimen. BTK inhibitors have demonstrated ideal therapeutic effects for the aforementioned patient types, and currently, a large number of patients have been treated with this type of therapy in clinical practice. However, the vast majority have been combined with R-CHOP-like regimens. There are no data reported on the combination of BTK inhibitors with the Pola regimen. Therefore, this study plans to assess the preliminary efficacy and safety of orelabrutinib in combination with the Pola-R-CHP regimen for the treatment of treatment-naive non-GCB diffuse large B-cell lymphoma (DLBCL). Enrolled patients will receive six cycles of orelabrutinib in combination with the Pola-R-CHP regimen, with each 21-day period being one cycle. At the end of the six cycles, an interim efficacy evaluation will be conducted. Patients with a response of CR or PR will receive an additional two cycles of orelabrutinib in combination with rituximab and undergo a final efficacy evaluation. Patients with a response of CR/PR after eight cycles of induction therapy will receive maintenance treatment with orelabrutinib for up to two years.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years old.
2. Diffuse large B-cell lymphoma (DLBCL) confirmed by tumor tissue pathology, with at least one measurable lesion.
3. Non-GCB.
4. No prior anti-tumor treatment.
5. ECOG score of 0-2.
6. Life expectancy of ≥6 months.
7. Voluntary written informed consent.

Exclusion Criteria:

1. Lymphoma involving the central nervous system or leptomeningeal metastasis.
2. Transformed lymphoma, that is, transformed from other types of lymphoma, such as follicular lymphoma, marginal zone lymphoma, chronic lymphocytic leukemia, or small B-cell lymphoma.
3. Primary mediastinal large B-cell lymphoma.
4. Burkitt lymphoma.
5. Laboratory values at screening (unless due to lymphoma):

   1. Neutrophils <1.5×10⁹/L;
   2. Platelets <75×10⁹/L;
   3. ALT or AST more than 2 times the upper limit of normal, ALP and bilirubin more than 1.5 times the upper limit of normal;
   4. Creatinine level more than 1.5 times the upper limit of normal.
6. Patients with psychiatric disorders or other known or suspected inability to fully comply with the study protocol.
7. Pregnant or breastfeeding women.
8. Known human immunodeficiency virus (HIV) infection, or active hepatitis B or C virus infection (positive result by polymerase chain reaction [PCR]). If the patient tests positive for HbsAg, HBV DNA testing is required. If HBV DNA <10³ IU/ml, the patient may be enrolled. If the patient tests negative for HbsAg but positive for HBcAb (regardless of HBsAb status), HBV DNA testing is also required. If HBV DNA <10³ IU/ml, the patient may be enrolled. If the patient tests positive for HCV antibody, HCV RNA is detected by PCR. If positive, the patient meets the exclusion criteria.
9. Need for continuous treatment with strong or moderate CYP3A inhibitors or CYP3A inducers.
10. Inability to swallow capsules or significant gastrointestinal disorders, such as malabsorption syndrome, bariatric surgery, inflammatory bowel disease, or partial or complete intestinal obstruction.
11. Other concurrent and uncontrolled medical conditions that the investigator believes will affect the patient's participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
2 years Progression free survival (2Y-PFS) | up to 2 years
  PFS is defined as the time from registration to the first occurrence of progression or relapse as assessed by the investigator, or death from any cause. PFS for patients without disease progression, relapse, or death will be censored at the time of the last tumor assessment

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to 8 months
  ORR is defined as the proportion of patients with a response of CR or PR
Complete Response Rate (CR) | up to 8 months
  The rate of patients who achieved complete response after treatment
overall survival (OS) | up to 3 years
  Overall survival is defined as the period from the induction registration to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China